CLINICAL TRIAL: NCT00757809
Title: A Blinded, Randomized, Multiple-Dose, Parallel Group Study to Characterize the Occurrence of Mild to Moderate Diarrhea After Administration of Neratinib Either 240-mg Once Daily or 120-mg Twice Daily for 14 Days to Healthy Subjects
Brief Title: Study Evaluating The Tolerability Of Multiple Doses Of HKI-272
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3144A1-1116
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- QD (Experimental): Once daily
  Interventions: Drug: neratinib
- BID (Experimental): Twice daily
  Interventions: Drug: neratinib

INTERVENTIONS:
Drug: neratinib — HKI-272

SUMMARY:
Study to investigate the occurence of diarrhea after either once daily or twice daily dosing for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female (non-child bearing potential) subjects
* Ages 18-50.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Occurence of diarrhea | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (2):
- United States (2):
  - Austin, Texas
  - Tacoma, Washington